CLINICAL TRIAL: NCT06132399
Title: Development and Validation of a Novel Virtual Reality Software for Improving Disability and Quality of Life in Patients With Stroke
Brief Title: Virtual Reality Software for Patients With Stroke
Acronym: RESET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government); European Union (Other)
Responsible Party: Principal Investigator, Alberto Soriano-Maldonado, PhD, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPP2021-008497
Record Dates: First submitted 2023-10-26; First posted 2023-11-15 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Stroke
Keywords: stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Commercial non-immersive virtual reality group (CVR) (Active Comparator): Nintendo Switch (Nintendo Co., Ltd, Kyoto, Japan).
  Interventions: Device: Nintendo Switch (Nintendo Co., Ltd, Kyoto, Japan)
- Gamified, fully immersive and stroke-specific virtual reality group (RESET) (Experimental): The RESET virtual reality software will be integrated in the META QUEST 3 glasses (Meta Platforms, San Francisco, CA, US).
  Interventions: Device: META QUEST 3 virtual reality glasses
- Usual care (UC) (Active Comparator): 3 session/week of 90 minutes of physical therapy and occupational therapy.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: META QUEST 3 virtual reality glasses — The RESET virtual reality software will be integrated into META QUEST 3 glasses (Meta Platforms, San Francisco, CA, US) by DYNAMICS.
  Arms: Gamified, fully immersive and stroke-specific virtual reality group (RESET)
Device: Nintendo Switch (Nintendo Co., Ltd, Kyoto, Japan) — This group will use the Nintendo Switch (Nintendo Co., Ltd, Kyoto, Japan) gaming system with the Sports package games.
  Arms: Commercial non-immersive virtual reality group (CVR)
Other: Usual care — The UC intervention consists of 3 sessions/week of 90' of physical therapy and occupational therapy conducted by a physiotherapist and an occupational therapist.
  Arms: Usual care (UC)

SUMMARY:
The goal os this clinical trial is to develop and validate a gamified, fully immersive, and stroke-specific virtual reality software to improve physical disability and quality of life in patients with stroke.

The main questions it aims to answer are:

* To assess the effects of a gamified, fully immersive and stroke-specific virtual reality 10-week intervention combined with usual care rehabilitation, compared to usual care rehabilitation alone and in combination with a commercially available VR system, on disability in patients with stroke.
* To assess the effects of a gamified, fully immersive and stroke-specific virtual reality intervention combined with usual care rehabilitation, compared to usual care rehabilitation alone and in combination with a commercially available virtual reality system, on quality of life, upper-body motor function, gross manual dexterity, handgrip strength, static and dynamic balance, and cognitive function in patients with stroke

DETAILED DESCRIPTION:
Stroke is the leading cause of long-term disability and ranks as the second most prevalent cause of mortality worldwide. According to data from the World Health Organization, since 2005, the global probability of a person experiencing a stroke has increased by 50 percent. It is expected that 1 in 4 individuals will face the risk of having a stroke in their lifetime. A stroke can result in significant loss of motor functions, communications abilities, weakness, or hemiparesis, leading to a diminished quality of life. Therefore, improving the rehabilitation process is evidently of paramount significance. Virtual reality has emerged as a novel strategy to improve neurological diseases; however, there is an absence of an immersive software designed specifically for stroke patients within a gamified environment. Therefore, the aim of RESET randomized controlled trial is to evaluate the effect of a gamified, fully immersive, and stroke-specific virtual reality software on disability in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Women and men with either an ischemic or hemorrhagic stroke
* Stroke between the last 7 to 14 days
* Functional independence before stroke (modified Rankin scale <3)
* Paresis of the lower extremity, upper extremity, or both, with a score ≤3 on the "motor arm" item of the National Institutes of Health Stroke Scale (NIHSS) scale
* Trunk control in seated and standing position
* Ability to understand basic instructions and to decide whether to sign informed consent

Exclusion Criteria:

* Moderate-severe aphasia that precludes understanding the required tasks
* Cognitive impairment that precludes cooperation with tasks
* Serious behavioral problems or mental disorders
* Lower extremity deep vein thrombosis, quadriplegia, neurodegenerative diseases, lower limb fractures, or recent myocardial infarction
* Vital organ (heart, lung, liver, kidney, etc.) failure, malignant tumor, or other unstable condition
* A history of cerebrovascular disease (if not fully resolved)
* Photosensitive epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Disability (The Barthel index) | Changes from baseline to weeks 13 and 26
  An ordinal scale used to measure performance in activities of daily living. It consists of 10 common activities, with eight of them representing activities related to personal care and 2 related to mobility. These are assessed for independence/dependence and scored via an arbitrary weighting system- the index yields a total score out of 100 - the higher the score, the lower degree of disability.

SECONDARY OUTCOMES:
Quality of life (NEWSQOL) | Changes from baseline to weeks 13 and 26
  The Newcastle Stroke-Specific Quality of Life Measure assess the specific health-related quality of life measure of 56 items grouped into 11 domains: feelings; ADL/self-care; cognition; mobility; emotion; sleep; interpersonal relationships; communication; pain/sensation; vision; and fatigue. Each item is rated in range 0 to 3, and they are not significant individually. The results of each domain are obtained by the sum of the scores of the items, and higher values indicate greater impact on quality of life.
Upper extremity motor function (Fugl-Meyer assessment of Upper Extremity) | Changes from baseline to weeks 13 and 26
  The test consists of 33 items that evaluate the movement, coordination and reflex action of the shoulder, elbow, forearm, wrist and hand. Each item is scored on a 3-point scale (0=cannot perform, 1=performs partially, 2=performs fully) and the total score ranges from a minimum of 0 (hemiplegia) to a maximum of 66 points.
Gross manual dexterity (The Box and Block Test) | Changes from baseline to weeks 13 and 26
  The participant is seated at a table, facing a rectangular box that is divided into two square compartments of equal dimension by means of a partition. A total of 150 colored, wooden cubes or blocks (2.5 cm) are placed in one compartment. The participant is instructed to move as many blocks as possible, one at a time, from one compartment to the other for 60 seconds. The score is the number of blocks moved from one compartment to the other during the trial time. The patient's hand must cross over the partition in order for a point to be given, and blocks that drop or bounce out of the second compartment onto the floor are still rewarded with a point. Multiple blocks carried over at the same time, count as a single point. Higher scores on the test indicate better gross manual dexterity.
Handgrip strength | Changes from baseline to weeks 13 and 26
  Digital dynamometry will be used to assess the muscular strength in kilograms of both the affected and non-affected upper extremities.Participants will execute the test three times with each hand and the best score will be used to calculate the average of the three repetitions. The non-paretic side will be used as a reference for the paretic side.
Lower extremity function (Berg Balance Scale) | Changes from baseline to weeks 13 and 26
  The Berg Balance Scale is a quantitative assessment of balance in older adults. The scale consists of 14 items requiring subjects to maintain positions or complete movement tasks (common to everyday life) of varying levels of difficulty. Items receive a score of 0-4 based on ability to meet the specific time and distance requirements of the test. 0 represents inability to complete the item and a 4 represents the ability to complete it independently.
Lower extremity function (Time Up and Go test) | Changes from baseline to weeks 13 and 26
  The Time Up and Go assesses the ability to perform sequential motor tasks relative to walking and turning. The test requires participants to stand up from a chair, walk a distance of 3 meters, turn around, walk back to the chair and seat by themselves in the minimum timeframe possible. The time taken to complete the test is registered.
Cognitive function | Changes from baseline to weeks 13 and 26
  The Montreal cognitive assessment, MoCA, consists of 10 simple questions or tasks related to cognitive function. Typically, these are grouped into the following cognitive domains: short term memory, visuospatial abilities, executive functions, attention, concentration, working memory, language, and orientation to time and place. The total score ranges 0-30. Higher scores indicating better cognitive performance.
Cognitive function | Changes from baseline to weeks 13 and 26
  The Trail-Making Test will be used to assess the executive function. Successful performance of this test requires letter and number recognition, mental flexibility, visual scanning, and motor function. The Part A consists of 25 circles with the numbers 1-25 written randomly in the circles. The participant is required to connect the circles with a pencil as quickly as possible (i.e. number one to number two, etc). The Part B of the test consists of 25 circles, 13 of them numbered 1 to 13 and, and 12 lettered A to L, randomly distributed over a page of paper. The participant is required to connect the circles with a pencil as quickly as possible, alternating between numbers and letters and taking both series in ascending sequence (i.e. 1, A, 2, B, 3, C…). The time taken to complete the task and the number of errors are recorded in seconds. Greater time indicates greater impairment.
Plasma concentrations of inflammatory markers | Changes from baseline to weeks 13 and 26
  Interleukin 2, 4, 6, 8, 10 (ng/mL)
BDNF quantification in blood | Changes from baseline to weeks 13 and 26
  Change in Brain-derived neurotrophic factor (ng/mL)
GDNF quantification in blood | Changes from baseline to weeks 13 and 26
  Change in Glial cell line-derived neurotrophic factor (ng/mL)
PACAP-38 quantification in blood | Changes from baseline to weeks 13 and 26
  Change in Pituitary Adenylate Cyclase-Activating Polypeptide-38 (ng/mL)
Plasma concentrations of inflammatory markers, quantification in blood | Changes from baseline to weeks 13 and 26
  Change in Tumor necrosis factor (TNF-alpha) (ng/mL)
IGF-1 quantification in blood | Changes from baseline to weeks 13 and 26
  Change in Insulin-Like Growth Factor-1 (ng/mL)
NGF quantification in blood | Changes from baseline to weeks 13 and 26
  Change in Nerve Growth Factor (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Soriano-Maldonado, PhD, Principal Investigator — Universidad de Almeria
Locations (4):
- Spain (4):
  - University of Almería, Almería, Almería
  - Torrecárdenas University Hospital, Almería
  - San Cecilio University Hospital, Granada
  - University of Granada, Granada

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data will be shared once the study is finalised and the main results are published. IPD can be obtained by contacting the responsible party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Two years (24 months) after the study completion.
Access Criteria: The PI must be contacted and a minimum number of co-authors from the research team must be included in any publication.

REFERENCES:
- [Derived] Hernandez-Martinez A, Fernandez-Escabias M, Amaya-Pascasio L, Carrilho-Candeias S, Ramos-Teodoro M, Gil-Rodriguez M, Orellana-Jaen A, Martinez-Rosales E, Ruiz-Gonzalez D, Esteban-Simon A, Castro-Ropero B, Del-Olmo-Iruela L, Lopez-Lopez MI, Ramos-Herrera AI, Fajardo-Rodriguez MF, Gomez-Garcia S, Rodriguez-Camacho M, Conde-Negri E, Rodriguez-Perez M, Marcos-Pardo PJ, Ruiz JR, Villegas-Rodriguez I, Amaro-Gahete FJ, Martinez-Sanchez P, Soriano-Maldonado A. Evaluation of the effects of a gamified, fully immersive and stroke-specific virtual reality intervention for improving disability and quality of life in patients with stroke in the subacute phase: study protocol of the RESET randomised trial. BMJ Open Sport Exerc Med. 2024 Aug 7;10(3):e002123. doi: 10.1136/bmjsem-2024-002123. eCollection 2024. PMID 39161559